CLINICAL TRIAL: NCT02657863
Title: Non-invasive Detection of Cancer DNA in Blood and Urine
Brief Title: Cancer DNA Detection in Blood and Urine
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Patrick C Walsh Prostate Cancer Research Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: J14106; IRB00043215 (Other: JHMIRB)
Record Dates: First submitted 2015-09-09; First posted 2016-01-18 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Urine Specimen Collection; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy volunteer: Normal volunteers will be enrolled and informed consent obtained per study guidelines as described. Urine and plasma will be collected from each of 30 subjects with no prior history of prostate or other cancers.
- Prostate cancer patients being treat with radiation therapy: Prostate cancer patients will be enrolled and informed consent obtained per study guidelines as described. We will collect urine and plasma samples from 25 consecutive men being treated with radiation therapy for high-risk prostate cancer prior to the onset of therapy.
- Prostate cancer patients being treated with radiation therapy: Prostate cancer patients will be enrolled and informed consent obtained per study guidelines as described. We will collect urine and plasma samples from 5 consecutive men being treated with radiation therapy for high-risk prostate cancer prior to initiation of androgen deprivation (week 0), again prior to initiation of radiotherapy (week 8), at the end of radiation therapy (week 16) and at 6 months and 12 months after the conclusion of radiation therapy.
  Interventions: Procedure: Urine collection and blood draw

INTERVENTIONS:
Procedure: Urine collection and blood draw
  Groups: Prostate cancer patients being treated with radiation therapy

SUMMARY:
This study is being conducted to collect and analyze biospecimens (blood and urine) and clinical data from patients with prostate cancer as well as healthy volunteers to better understand the differences between cancer cells and normal tissues with the goal of developing a better way to detect and track the treatment of prostate cancer.

* These samples are being collected to conduct research to accomplish the goal of improving cancer therapies, biomarkers, and hopefully lead to more effective treatment of prostate cancer.
* The samples that you are providing as a patient with prostate cancer will be used in future research.
* Your biospecimens will be compared to the cancer and normal volunteer specimens from other participants to understand genetic differences between normal and cancer cells. Genetic material, including DNA and RNA, will be obtained from samples, stored, and used for evaluation.
* Clinical information and samples will be collected and stored for ongoing research. This is a necessity because improved diagnosis, prognosis and treatment of cancer in the future depend upon the ongoing analysis of basic research findings and clinical outcomes. This type of research may improve the lives of future patients with cancer.

Men between the ages of 18 and 100 with a diagnosis of cancer undergoing standard therapy with radiation may join.

DETAILED DESCRIPTION:
The American Cancer Society estimates that approximately 29,480 men will die of prostate cancer in the United States in 2014. Many of these men were initially diagnosed with aggressive prostate cancer (so-called "high risk" prostate cancer), often with cancer that extended beyond the prostate gland itself or was of a high Gleason score, or was associated with a Prostate Specific Antigen [PSA] level > 20 ng/ml. In contrast to the more favorable outcomes in men with low and intermediate risk disease, nearly 50% of men with high-risk prostate cancer will have a recurrence of their cancer despite a complete course of treatment. One of the mainstays of care for men with high-risk prostate cancer is a combination of radiation therapy and hormone suppression (more appropriately called androgen deprivation [ADT]). Despite advances, a clear need exists for improved clinical management of high risk disease.

One of the challenges in the overall management of men with high risk prostate cancer is the lack of a reliable test allowing clinicians to monitor tumor response both during and after radiation therapy. The commonly used marker, prostate specific antigen (PSA), is less useful in men receiving ADT. In these men, the PSA is level is strongly suppressed by the ADT and is a less reliable surrogate for detecting active tumor. Importantly, ADT is given both during and for up to 3 years following radiation therapy, limiting the utility of PSA testing for an extended period of time during which the window for curative therapies may close. The development of an accurate, noninvasive monitoring test is needed, to guide early implementation of salvage strategies aimed at increasing the proportion of patients cured of their disease.

Prior research from our group and several others has demonstrated that prostate cancers nearly universally harbor stable, cancer-specific changes (modifications) of the DNA. Furthermore, published studies have shown that this modified (methylated) DNA can be readily detected in urine and blood specimens from men with primary prostate cancer.

Investigators hypothesize that large scale assessment of cancer-specific DNA changes and rearrangements in the urine and plasma of prostate cancer patients using technology developed by our group (qMBD-seq), will allow for more informative and accurate tracking of disease burden and therapeutic response in men receiving radiation therapy and ADT for high-risk prostate cancer.

Investigators have two straightforward primary objectives for this pilot study. First we will establish the background levels of modified DNA in individuals with no history of prostate cancer. Second, investigators will quantify cancer-specific methylated DNA in men with known high risk prostate cancer. Investigators will begin by collecting urine and plasma specimens from normal volunteers. In parallel investigators will collect specimens for quantitation of cancer-specific DNA modifications in men with known high-risk prostate cancer receiving standard treatment in the Department of Radiation Oncology. Patient samples will be collected at multiple time points before, during, and after radiation treatment and then will be subjected to careful DNA sequencing and analysis. This will allow investigators to simultaneously characterize and quantify prostate cancer specific DNA occurring anywhere in the genome, thereby allowing investigators to predict which patients have prostate cancer still present in their body after treatment even if the PSA is very low or undetectable. If successful, this project will be an important first step in the development of a noninvasive test to track disease burden and therapeutic response during and after radiation therapy for high-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male older than or equal to 18 years of age, but not older than 100 years of age.
2. Signed informed consent prior to initiation of any study-related procedures.
3. Minorities are included in this protocol.
4. Signed informed consent prior to initiation of any study-related

Exclusion Criteria:

1. It is the enrolling study physician's discretion to decide if a patient is not fit enough to undergo procedures outlined in this protocol.
2. Persons who are incarcerated are not eligible to participate.
3. Women are not eligible.
4. Persons incapable of providing informed consent are not eligible.
5. Any person with a personal history of prior malignancy is not eligible
6. Persons with an inherited cancer syndrome or a medical history suggestive of an inherited cancer syndrome are not eligible.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and men with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Healthy volunteer baseline | day 1
  Establish the background reference range for cancer specific DNA methylation and structural alterations in urine and plasma from normal individuals.
DNA alterations in blood and urine during radiation therapy | blood and urine draw at baseline, week 8 of treatment and then at week 16 of treatment
  Examine cancer-specific DNA methylation and structural alterations in urine and plasma during and after fractionated radiation therapy for men with high-risk prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore DeWeese, M.D., Principal Investigator — Johns Hopkin SKCCC
Locations (1):
- Johns Hopkins SKCCC, Baltimore, Maryland, United States